CLINICAL TRIAL: NCT00467077
Title: Phase II Trial of ZD1839 (IRESSA®) and Pegylated Interferon Alfa 2b (PEG-Intron™) in Unresectable or Metastatic Renal Cell Carcinoma
Brief Title: Gefitinib and PEG-Interferon Alfa-2b in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol was closed due to slow accrual.
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540598; P30CA093373 (NIH); CCC-PHII-40; ZENECA-AZ1839US/0227; UCD-200412338-4; UCD-ZD1839
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; stage III renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — peginterferon alfa-2b; Gefitinib

ARMS (1):
- Gefitinib and PEG-IFNa Treatment (Experimental): Gefitinib administered at a dose of 250 mg orally once daily for 12 weeks. PEG-IFNa at 4.0 µg/kg/wk administered subcutaneously once weekly for 6 weeks (cycle repeated once for a total of 2 cycles).
  Interventions: Biological: PEG-interferon alfa-2b; Drug: gefitinib

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — PEG-Interferon will be administered subcutaneously (sq) once weekly for 6 weeks
Drug: gefitinib — ZD1839 will be administered at a dose of 250 mg orally once daily,

SUMMARY:
RATIONALE: Gefitinib may stop the growth of kidney cancer by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. PEG-interferon alfa-2b may interfere with the growth of tumor cells and slow the growth of kidney cancer. Giving gefitinib together with PEG-interferon alfa-2b may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gefitinib together with PEG-interferon alfa-2b works in treating patients with unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month progression-free survival of patients with unresectable or metastatic renal cell carcinoma treated with gefitinib and PEG-interferon alfa-2b.

Secondary

* Determine the response rate (by RECIST criteria), duration of response, time to treatment failure, and overall survival of patients treated with this regimen.
* Assess toxicity and tolerability of this regimen in these patients.
* Determine the pre-treatment expression of the von Hippel-Lindau (VHL) protein, the epidermal growth factor receptor (EGFR), and p27, and correlate with response to treatment.
* Determine post-treatment alteration of EGFR and p27 expression in patients with tumors accessible for serial biopsy.
* Assess changes in EGFR levels in buccal epithelial cells in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once daily and PEG-interferon alfa-2b subcutaneously once weekly in weeks 1-6. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with a partial response or stable disease after completion of course 2 continue to receive gefitinib alone as above in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma

  * Metastatic or advanced/unresectable disease
* Measurable or nonmeasurable disease as defined by RECIST criteria
* No uncontrolled brain metastases

  * Patients with adequately treated brain metastases who are not taking anticonvulsants and corticosteroids may be eligible

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,500/mm³
* Platelet count ≥ 100,000/mm³
* Absolute granulocyte count ≥ 1,500/mm³
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 50 mL/min
* Bilirubin ≤ 1.5 mg/dL
* AST ≤ 2 times upper limit of normal (ULN)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or adequately treated stage I or II cancer from which the patient is currently in complete remission
* No known severe hypersensitivity to gefitinib or its excipients
* No incomplete healing from previous oncologic or other major surgery
* No unresolved chronic toxicity > grade 2 from previous anticancer therapy (except alopecia and anemia)
* No evidence of clinically active interstitial lung disease

  * Patients with chronic stable radiographic changes who are asymptomatic are eligible
* No evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* No other significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior nonapproved or investigational drugs
* More than 6 weeks since prior aldesleukin or interferon and recovered
* At least 3 weeks since prior radiotherapy
* No prior gefitinib
* Prior chemotherapy or biological therapy allowed
* Prior or concurrent bisphosphonate therapy for bone metastases allowed
* No concurrent phenytoin, carbamazepine, rifampin, barbiturates, phenobarbital, or Hypericum perforatum (St. John's wort)
* No other concurrent agents specifically designed to inhibit the epidermal growth factor receptor (EGFR)
* No concurrent radiotherapy to measurable lesions

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California

REFERENCES:
- [Derived] Shek D, Longmate J, Quinn DI, Margolin KA, Twardowski P, Gandara DR, Frankel P, Pan CX, Lara PN Jr. A phase II trial of gefitinib and pegylated IFNalpha in previously treated renal cell carcinoma. Int J Clin Oncol. 2011 Oct;16(5):494-9. doi: 10.1007/s10147-011-0212-8. Epub 2011 Mar 23. PMID 21431345

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gefitinib and PEG-IFNa Treatment
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib and PEG-IFNa Treatment
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 60 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Six-month Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-target lesions
Time Frame: From the date treatment started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gefitinib and PEG-IFNa Treatment
Number analyzed (Participants) | 21
percentage of participants | 29 [15 to 56]

2. Secondary Outcome: Number of Participants With Overall Response as Measured by RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response = CR + PR
Time Frame: After 2 cycles of treatment, up to 2 years.
Measure: Number; unit: participants
Arm/Group | Gefitinib and PEG-IFNa Treatment
Number analyzed (Participants) | 21
participants | 2

3. Secondary Outcome: Progression-Free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Until disease progression, up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib and PEG-IFNa Treatment
Number analyzed (Participants) | 21
Months | 5.2 [3.0 to 10.1]

4. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib and PEG-IFNa Treatment
Number analyzed (Participants) | 21
Months | 13.6 [10.3 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 38 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Arm 1: Gefitinib administered at a dose of 250 mg orally once daily for 12 weeks. PEG-IFNa at 4.0 µg/kg/wk administered subcutaneously once weekly for 6 weeks (cycle repeated once for a total of 2 cycles).
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=21)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Leukopenia (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (63)
Cardiac disorder (Cardiac disorders) | 1 (3)
Palpitations (Cardiac disorders) | 1 (1)
Conjunctival disorder (Eye disorders) | 1 (6)
Dry eye syndrome (Eye disorders) | 1 (3)
Eye disorder (Eye disorders) | 1 (1)
Eyelid function disorder (Eye disorders) | 2 (11)
Retinopathy (Eye disorders) | 1 (3)
Vision blurred (Eye disorders) | 2 (3)
Watering eyes (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (9)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (28)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (21)
Vomiting (Gastrointestinal disorders) | 8 (10)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 7 (7)
Edema limbs (General disorders) | 2 (12)
Fatigue (General disorders) | 17 (48)
Fever (General disorders) | 2 (2)
Flu-like symptoms (General disorders) | 1 (1)
Gait abnormal (General disorders) | 1 (2)
General symptom (General disorders) | 1 (2)
Injection site reaction (General disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Eye infection (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 2 (2)
Nail infection (Infections and infestations) | 1 (3)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (3)
Scrotal infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (15)
Alkaline phosphatase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 10 (22)
Bilirubin increased (Investigations) | 2 (9)
Creatinine increased (Investigations) | 8 (34)
Hyperbilirubinemia (Investigations) | 3 (4)
INR increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 5 (10)
Leukopenia (Investigations) | 11 (18)
Lymphocyte count decreased (Investigations) | 4 (10)
Lymphopenia (Investigations) | 3 (5)
Neutrophil count decreased (Investigations) | 10 (16)
Platelet count decreased (Investigations) | 6 (9)
Weight loss (Investigations) | 6 (18)
Anorexia (Metabolism and nutrition disorders) | 13 (29)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (11)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (36)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (16)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (10)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (9)
Dizziness (Nervous system disorders) | 5 (9)
Headache (Nervous system disorders) | 2 (8)
Memory impairment (Nervous system disorders) | 2 (14)
Peripheral motor neuropathy (Nervous system disorders) | 1 (3)
Sinus pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (19)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 4 (7)
Depression (Psychiatric disorders) | 5 (26)
Euphoria (Psychiatric disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 3 (4)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (4)
Urinary retention (Renal and urinary disorders) | 1 (3)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (16)
Acne (Skin and subcutaneous tissue disorders) | 5 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (19)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (5)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (19)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (28)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Protocol was closed prior to the second stage of accrual (pegged at n = 24) due to slow accrual. The reason for the slow accrual was likely the availability of several new Food and Drug Administration approved targeted agents during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less